CLINICAL TRIAL: NCT00964223
Title: A Single-blind, Randomized, Comparative Split-face Study Evaluating the Tolerability of Clindamycin and Benzoyl Peroxide Gel to Benzoyl Peroxide/Adapalene Gel in the Treatment of Acne Vulgaris.
Brief Title: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Facial Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114547
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duac gel (Experimental): Subjects will apply Duac gel once a day to one-half of their face and and apply Epiduo gel on the other side of their face once daily for the first 2 weeks.
  Interventions: Drug: Clindamycin and benzoyl peroxide gel (Duac® Topical Gel)
- Epiduo gel (Active Comparator): Subjects will apply Duac gel once a day to one-half of their face and and apply Epiduo gel on the other side of their face once daily for the first 2 weeks.
  Interventions: Drug: benzoyl peroxide and adapalene gel (EPIDUO™ Gel)

INTERVENTIONS:
Drug: Clindamycin and benzoyl peroxide gel (Duac® Topical Gel) — Subjects will apply Duac(clindamycin and benzoyl peroxide) gel to one-half of their face and and apply Epiduo (benzoyl peroxide/adapalene) gel on the other side of their face once a day for the first 2 weeks. Starting at week 2, subjects will apply Duac (benzoyl peroxide/clindamycin gel) to the entire face for an additional 6 weeks.
  Other Names: Duac® Topical Gel
  Arms: Duac gel
Drug: benzoyl peroxide and adapalene gel (EPIDUO™ Gel) — Subjects will apply Duac(clindamycin and benzoyl peroxide) gel to one-half of their face and and apply Epiduo (benzoyl peroxide/adapalene) gel on the other side of their face once a day for the first 2 weeks. Starting at week 2, subjects will apply Duac (benzoyl peroxide/clindamycin gel) to the entire face for an additional 6 weeks.
  Other Names: EPIDUO™ Gel
  Arms: Epiduo gel

SUMMARY:
Multi-center, single-blind, randomized, comparative, split-face study. The duration of the study is 8 weeks. Commencing at baseline, subjects will apply once daily both clindamycin and benzoyl peroxide gel and benzoyl peroxide/adapalene gel in a bilateral split-face fashion (allocation to left and right side randomly assigned) for an initial 2 weeks. After visit 3, subjects will commence application of clindamycin and benzoyl peroxide gel to the entire face for an additional 6 weeks.

DETAILED DESCRIPTION:
Multi-center, single-blind, randomized, comparative, split-face study. The duration of the study is 8 weeks and consists of a baseline visit and visits at weeks 1, 2, 5 and 8. Commencing at baseline, subjects will apply once daily both clindamycin and benzoyl peroxide gel and benzoyl peroxide/adapalene gel in a bilateral split-face fashion (allocation to left and right side randomly assigned) for an initial 2 weeks. After visit 3 subjects will commence application of clindamycin and benzoyl peroxide gel to the entire face for an additional 6 weeks.

Blinding This is an investigator-blinded study; therefore, subjects and study-center staff will not be blinded to study treatment allocation (ie, left vs. right side application). During the first 2 weeks, the investigator will be unaware of which study product is being used on either side of the face. Subjects and study-center staff will be instructed not to reveal study treatment allocation to the investigator. Subjects will be instructed not to use study product in the presence of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age, in good general health with documented diagnosis of facial acne vulgaris.
* Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product.
* Subjects willing to follow therapeutic instructions including avoidance of any other topical facial or systemic acne therapy during the conduct of the study.
* Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed.

Exclusion Criteria:

* Female subjects who are pregnant, trying to become pregnant or breastfeeding.
* Subjects who have any clinically relevant finding at their baseline physical examination or medical history such as severe systemic diseases, diseases of the facial skin, other than acne vulgaris.
* Facial hair that may obscure the accurate assessment of acne grade.
* History or presence of regional enteritis or inflammatory bowel disease (e.g., ulcerative colitis, pseudomembranous colitis, chronic diarrhea, or a history of antibiotic-associated colitis) or similar symptoms.
* Use of topical antibiotics on the face and systemic antibiotics within the past 2 and 4 weeks, respectively.
* Use of topical corticosteroids on the face or systemic corticosteroids within the past 4 weeks. Use of inhaled, intra-articular or intra-lesional (other than for facial acne lesions) steroids is acceptable.
* Use of systemic retinoids within the past 6 months.
* Concurrent use of drugs known to be photosensitizers (e.g., thiazides, tetracyclines, fluoroquinolones, phenothiazines, sulfonamides) because of the possibility of increased phototoxicity.
* Concomitant use of neuromuscular blocking agents. Clindamycin has neuromuscular blocking activities, which may enhance the action of other neuromuscular blocking agents.
* Use of topical anti-acne medications within the past 2 weeks.
* Use of any investigational drugs or treatments during the study or within 4 weeks of the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Aesthetics, Skin Care & Dermasurgery, Rockville, Maryland
  - Grekin Skin Institute, Warren, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gonzalez P, Vila R, Cirigliano M. The tolerability profile of clindamycin 1%/benzoyl peroxide 5% gel vs. adapalene 0.1%/benzoyl peroxide 2.5% gel for facial acne: results of a randomized, single-blind, split-face study. J Cosmet Dermatol. 2012 Dec;11(4):251-60. doi: 10.1111/jocd.12013. PMID 23174047
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114547 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research centers
Groups:
- All Study Participants: Commencing at baseline, subjects will apply once daily both clindamycin and benzoyl peroxide and benzoyl peroxide/adapalene gel in a bilateral split-face fashion (allocation to left and right side randomly assigned) for an initial 2 weeks. After visit 3, subjects will commence application of clindamycin and benzoyl peroxide gel to the entire face for an additional 6 weeks.
Period: Split Face Treatment (Weeks 1 and 2)
Arm/Group | All Study Participants
Started | 28
Completed | 28
Not Completed | 0
Period: Full Face Treatment (Weeks 5 and 8)
Arm/Group | All Study Participants
Started | 28
Completed | 27
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  Black or African American | 11
  White | 15
Region of Enrollment [Number; unit: participants]
  United States | 28
Investigators Static Global Assessment (ISGA) [Number; unit: Participants] — Patients with the following ISGA grades were eligible for enrollment on this study: 0, Clear: clear skin with no inflammatory lesions (IL) or non-inflammatory lesions (NIL); 1, Almost clear: rare NIL with no more than one small IL; 2, Mild: some NIL with no more than a few IL (papules/pustules only, no nodular lesions); 3, Moderate: up to many NIL and may have some IL, but no more than one small nodular lesion; 4, Severe: up to many NIL and IL, but no more than a few small nodular lesions; 5, Very severe: many NIL and IL and more than a few nodular lesions. May have cystic lesions.
  Participants
    Mild | 2
    Moderate | 20
    Severe | 6
Inflammatory Acne Lesion Count [Mean (Standard Deviation); unit: Inflammatory Lesion] — Inflammatory acne lesion count at baseline (number of pustules and papules).
  Inflammatory Lesion | 21.5 (9.3)
Non-Inflammatory Acne Lesion Count [Mean (Standard Deviation); unit: Non-Inflammatory lesion] — Non-Inflammatory acne lesion count at baseline (number of whiteheads and blackheads)
  Non-Inflammatory lesion | 33.0 (24.7)
Total Acne Lesion Count [Mean (Standard Deviation); unit: Acne lesions] — Total acne lesion count (includes inflammatory and non-inflammatory lesions)
  Acne lesions | 54.5 (27.1)

OUTCOME MEASURES:

1. Primary Outcome: Skin Dryness Score
Description: Investigator assessment of tolerability (skin dryness) on the face. Erythema, peeling, and dryness were graded using the following Investigator Assessment of Tolerability scale: 0, None; 1, Slight; 2, Moderate; 3, Intense.
Time Frame: Week 1, Week 2
Population: Intent-to-Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Duac Gel; Epiduo Gel: Starting at baseline, subjects will apply once daily both clindamycin and benzoyl peroxide and benzoyl peroxide/adapalene gel in a bilateral split-face fashion (allocation to left and right side randomly assigned) for an initial 2 weeks. After visit 3, subjects will commence application of clindamycin and benzoyl peroxide gel to the entire face for an additional 6 weeks.
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 0.15 (0.37) | 0.46 (0.71)
  Week 2 | 0.14 (0.36) | 0.29 (0.53)

2. Primary Outcome: Skin Peeling Score
Description: Investigator assessment of tolerability (skin peeling) on the face. Erythema, peeling, and dryness were graded using the following Investigator Assessment of Tolerability scale: 0, None; 1, Slight; 2, Moderate; Intense, 3.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 0.15 (0.37) | 0.54 (0.71)
  Week 2 | 0.18 (0.39) | 0.21 (0.50)

3. Primary Outcome: Irritant/Allergic Contact Dermatitis Score
Description: Signs and symptoms of tolerability (erythema, peeling, dryness, and irritant/allergic contact dermatitis) on the face.
  Erythema,peeling, and dryness were graded using the following scale:
  0 None
  1. Slight
  2. Moderate
  3. Intense
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 0.00 (0.00) | 0.15 (0.46)
  Week 2 | 0.00 (0.00) | 0.00 (0.00)

4. Primary Outcome: Erythema (Redness) Score
Description: Investigator assessment of tolerability (irritant/allergic contact dermatitis) on the face. Erythema, peeling, and dryness were graded using the following Investigator Assessment of Tolerability scale: 0, None; 1, Slight; 2, Moderate; 3, Intense.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 0.27 (0.53) | 0.58 (0.81)
  Week 2 | 0.18 (0.39) | 0.36 (0.49)

5. Secondary Outcome: Erythema (Redness) Score
Description: Investigator assessment of tolerability (erythema) on the face. Erythema, peeling, and dryness were graded using the following Investigator Assessment of Tolerability scale: 0, None; 1, Slight; 2, Moderate; 3, Intense.
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Week 5 | 0.26 (0.53)
  Week 8 | 0.19 (0.40)

6. Secondary Outcome: Skin Dryness Score
Description: as for outcome 1
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Week 5 | 0.15 (0.46)
  Week 8 | 0.00 (0.00)

7. Secondary Outcome: Skin Peeling Score
Description: Investigator assessment of tolerability (skin peeling) on the face. Erythema, peeling, and dryness were graded using the following Investigator Assessment of Tolerability scale: 0, None; 1, Slight; 2, Moderate; 3, Intense.
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Week 5 | 0.00 (0.00)
  Week 8 | 0.00 (0.00)

8. Secondary Outcome: Irritant/Allergic Contact Dermatitis Score
Description: Investigator assessment of tolerability (contact dermatitis) on the face. Erythema, peeling, and dryness were graded using the following Investigator Assessment of Tolerability scale: 0, None; 1, Slight; 2, Moderate; 3, Intense.
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Week 5 | 0.04 (0.19)
  Week 8 | 0.00 (0.00)

9. Secondary Outcome: Investigator Static Global Assessment Score
Description: ISGA is evaluated using the following scale: 0, clear, clear skin with no lesions; 1, almost clear, rare non-inflammatory lesions; 2, mild, some non-inflammatory lesions with no more than a few inflammatory lesions but no nodular lesions; 3, moderate, up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than 1 small nodular lesion; 4, severe, up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions; 5, very severe, many non-inflammatory and inflammatory lesions and more than a few nodular lesions. May have cystic lesions.
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Week 5 | 2.63 (0.93)
  Week 8 | 2.15 (1.03)

10. Secondary Outcome: Inflammatory Acne Lesion Counts
Description: Total number of inflammatory acne lesions (pustules, papules) at each timepoint.
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: inflammatory acne lesions
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
inflammatory acne lesions
  Week 5 | 8.44 (7.57)
  Week 8 | 7.00 (9.03)

11. Secondary Outcome: Non-Inflammatory Acne Lesion Counts
Description: Total number of non-inflammatory acne lesions (whiteheads and blackheads) at each timepoint.
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: non-inflammatory acne lesions
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
non-inflammatory acne lesions
  Week 5 | 14.37 (11.20)
  Week 8 | 10.81 (8.88)

12. Secondary Outcome: Total Acne Lesion Counts
Description: Total acne lesion counts - includes both inflammatory acne lesions (pustules, papules), noninflammatory lesions (whiteheads and blackheads),
Time Frame: Week 5, Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: total acne lesions
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
total acne lesions
  Week 5 | 22.81 (14.87)
  Week 8 | 17.81 (14.04)

13. Secondary Outcome: Skindex-29 Quality of Life Questionnaire - Symptomatic Domain
Description: Skindex-29 Quality of Life (QoL) Questionnaire used in dermatological disease consisting of 29 questions covering: burden of symptoms, functioning and emotional domains, with a five-point scale from: "never" to "all the time", higher scores for each domain indicate worse effects on QoL. Scores range from 0 to 100. Higher scores indicate worse QoL for that domain.
Time Frame: Baseline, and Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Baseline | 28.10 (17.01)
  Week 8 | 21.72 (11.60)

14. Secondary Outcome: Skindex-29 Quality of Life Questionnaire - Emotional Domain
Description: Skindex-29 Quality of Life (QoL)Questionnaire used in dermatological disease consisting of 29 questions covering: burden of symptoms, functioning and emotional domains, with a five-point scale from: "never" to "all the time", higher scores for each domain indicate worse effects on QoL. Scores range from 0 to 100. Higher scores indicate worse QoL for that domain.
Time Frame: Baseline, and Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Baseline | 44.29 (28.03)
  Week 8 | 35.37 (26.03)

15. Secondary Outcome: Skindex-29 Quality of Life Questionnaire - Functional Domain
Description: as for outcome 14
Time Frame: Baseline, and Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Baseline | 14.06 (13.41)
  Week 8 | 9.10 (10.39)

16. Secondary Outcome: Skindex-29 Quality of Life Questionnaire - Global Score
Description: Skindex-29 Quality of Life (QoL)Questionnaire used in dermatological disease consisting of 29 questions covering: burden of symptoms, functioning and emotional domains, with a five-point scale from: "never" to "all the time", higher scores for each domain indicate worse effects on QoL. The Global Score ranges from 0 to 100. Higher scores indicate worse QoL for that domain.
Time Frame: Baseline, and Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale
  Baseline | 14.06 (13.41)
  Week 8 | 9.10 (10.39)

17. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Redness
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 0, none; 1, very minimal; 2, mild; 3, moderate; 4, severe; 5, very severe.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 1.12 (1.24) | 1.54 (1.36)
  Week 2 | 0.78 (0.80) | 1.00 (0.89)

18. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Redness
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 0, none; 1, very minimal; 2, mild; 3, moderate; 4, severe; 5, very severe.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 1.00 (1.14)

19. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Dryness
Description: as for outcome 17
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 1.42 (1.36) | 1.88 (1.82)
  Week 2 | 1.31 (1.23) | 1.58 (1.27)

20. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Dryness
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 1.22 (1.12)

21. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Burning
Description: as for outcome 17
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 1.12 (1.24) | 1.96 (1.61)
  Week 2 | 0.73 (0.92) | 1.11 (1.31)

22. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Burning
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 0.63 (0.93)

23. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Itching
Description: as for outcome 17
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 1.19 (1.13) | 1.42 (1.30)
  Week 2 | 0.81 (1.02) | 1.19 (1.27)

24. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Itching
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 0.63 (1.01)

25. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Scaling
Description: as for outcome 17
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 0.77 (1.07) | 1.15 (1.32)
  Week 2 | 0.69 (0.93) | 1.00 (1.17)

26. Secondary Outcome: Product Acceptability and Preference Questionnaire - Severity of Scaling
Description: as for outcome 18
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 0.78 (1.28)

27. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Application of Product
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 1, very easy; 2, easy; 3, neutral; 4, difficult; 5, very difficult.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 1.46 (0.58) | 1.50 (0.71)
  Week 2 | 1.43 (0.50) | 1.50 (0.84)

28. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Application of Product
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, very easy; 2, easy; 3, neutral; 4, difficult; 5, very difficult.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 1.26 (0.45)

29. Secondary Outcome: Product Acceptability and Preference Questionnaire - Comfort of Skin
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 1, very comfortable; 2, comfortable; 3, somewhat comfortable; 4, somewhat uncomfortable; 5, uncomfortable.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 2.38 (0.94) | 2.58 (1.24)
  Week 2 | 2.00 (0.86) | 2.25 (1.14)

30. Secondary Outcome: Product Acceptability and Preference Questionnaire - Comfort of Skin
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, very comfortable; 2, comfortable; 3, somewhat comfortable; 4, somewhat uncomfortable; 5, uncomfortable.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 1.78 (0.85)

31. Secondary Outcome: Product Acceptability and Preference Questionnaire - Which Study Product is Subject More Satisfied With?
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 1 and week 2 asking which study product they were more satisfied with: Duac or Epiduo.
Time Frame: Week 1, Week 2
Population: ITT. Some participants missed a visit and therefore were not included in the number of participants analyzed for that visit.
Measure: Number; unit: Participants
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Participants
  Week 1 | 17 | 8
  Week 2 | 12 | 15

32. Secondary Outcome: Product Acceptability and Preference Questionnaire - Comparison of Study Products to Products Used in the Past
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, more satisfied; 2, somewhat more satisfied; 3, neither satisfied or dissatisfied; 4, more satisfied; 5, more dissatisfied.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 1.93 (1.24)

33. Secondary Outcome: Product Acceptability and Preference Questionnaire - Decrease of Acne Breakouts by Study Products
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 1, highly favorable; 2, favorable; 3, neutral; 4, unfavorable; 5, highly unfavorable.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 2.27 (0.78) | 2.27 (0.72)
  Week 2 | 2.14 (0.80) | 2.07 (0.81)

34. Secondary Outcome: Product Acceptability and Preference Questionnaire - Decrease of Acne Breakouts by Study Products
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, highly favorable; 2, favorable; 3, neutral; 4, unfavorable; 5, highly unfavorable.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 2.07 (1.14)

35. Secondary Outcome: Product Acceptability and Preference Questionnaire - Compliance
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 0, non-compliant (< 50% of the week); 1, mostly compliant (50-79%); 2, very compliant (80-100%).
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 1.96 (0.20) | 1.93 (0.20)
  Week 2 | 1.93 (0.26) | 1.93 (0.26)

36. Secondary Outcome: Product Acceptability and Preference Questionnaire - Compliance
Description: Subject response to question regarding use of the product every day or not at week 8 time point answering Yes or No
Time Frame: Week 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Participants
  Yes | 24
  No | 3

37. Secondary Outcome: Product Acceptability and Preference Questionnaire - Feeling of Hydrated and Moisturized Skin
Description: Subject response to question: did you feel that your skin was hydrated and moisturized while you on your study product? (Yes or No).
Time Frame: Week 1, Week 2
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Participants
  Week 1 - Yes | 18 | 16
  Week 1 - No | 8 | 10
  Week 2 - Yes | 19 | 18
  Week 2 - No | 8 | 9

38. Secondary Outcome: Product Acceptability and Preference Questionnaire - Feeling of Hydrated and Moisturized Skin
Description: as for outcome 37
Time Frame: Week 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Participants
  Yes | 24
  No | 3

39. Secondary Outcome: Product Acceptability and Preference Questionnaire - Use of Study Product if Choice to Continue Acne Treatment
Description: Subject response to the following question: If you were to choose to continue treatment for your acne, which treatment would you choose? (Yes or No).
Time Frame: Week 1, Week 2
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Participants
  Week 1 - Yes | 19 | 15
  Week 1 - No | 5 | 10
  Week 2 - Yes | 16 | 18
  Week 2 - No | 10 | 9

40. Secondary Outcome: Product Acceptability and Preference Questionnaire - Use of Study Product if Choice to Continue Acne Treatment
Description: as for outcome 39
Time Frame: Week 8
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Participants
  Yes | 20
  No | 7

41. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Use With Make-Up
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 0, not applicable; 1, very easy; 2, easy; 3, neutral; 4, difficult.
Time Frame: Week 1, Week 2
Population: ITT. All participants were asked to respond to the questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 2.31 (1.11) | 2.38 (1.12)
  Week 2 | 1.59 (0.87) | 1.59 (0.87)

42. Secondary Outcome: Product Acceptability and Preference Questionnaire - Ease of Use With Make-Up
Description: Measure Description Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 0, not applicable; 1, very easy; 2, easy; 3, neutral; 4, difficult.
Time Frame: Week 8
Population: ITT. All participants were asked to respond to the questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 1.89 (0.96)

43. Secondary Outcome: Product Acceptability and Preference Questionnaire - Overall Satisfaction of Study Product
Description: Product Acceptability and Preference Questionnaire was completed by the subject at weeks 1 and 2 using the following scale: 1, very satisfied; 2, satisfied; 3, neutral; 4, unsatisfied; 5, very unsatisfied.
Time Frame: Week 1, Week 2
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel | Epiduo Gel
Number analyzed (Participants) | 28 | 28
Units on a scale
  Week 1 | 2.04 (0.92) | 2.19 (1.06)
  Week 2 | 2.21 (1.17) | 2.32 (1.16)

44. Secondary Outcome: Product Acceptability and Preference Questionnaire - Overall Satisfaction of Study Product
Description: Product Acceptability and Preference Questionnaire was completed by the subject at week 8 using the following scale: 1, very satisfied; 2, satisfied; 3, neutral; 4, unsatisfied; 5, very unsatisfied.
Time Frame: Week 8
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duac Gel
Number analyzed (Participants) | 28
Units on a scale | 2.52 (1.37)

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.